CLINICAL TRIAL: NCT01464762
Title: Early Access of TMC207 in Combination With Other Anti-Tuberculosis (TB) Drugs in Subjects With Extensively Drug Resistant (XDR) or Pre-XDR Pulmonary Tuberculosis
Brief Title: Early Access of TMC207 in Patients With Extensively Drug Resistant or Pre-XDR Pulmonary Tuberculosis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017233; TMC207TBC3001 (Other: Janssen Infectious Diseases BVBA); 2010-021125-12 (EudraCT Number)
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TMC207TBC3001; TMC207; Early access; TB; Drug resistant; Multi drug-resistant; Extensively drug-resistant
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline

INTERVENTIONS:
Drug: TMC207 — 400mg once daily by mouth for 2 weeks followed by 200mg by mouth three times per week for 22 weeks + individualized background of antibacterial drugs

SUMMARY:
The purpose of this is a study to provide early access of TMC207 to patients with pulmonary infection due to strains of Mycobacterium tuberculosis (M. tuberculosis) with resistance to isoniazid (INH), rifampin (RMP), and to a fluoroquinolone (FQ) and/or injectable second line tuberculosis (TB) drug (kanamycin, amikacin, or capreomycin) and who are unable/ineligible to participate in any other TMC207 study. In addition, information on safety and tolerability of TMC207 in combination with anti-TB drugs will be assessed and the results of microbiology assessments which are recommended to be performed during the early access study will be collected.

DETAILED DESCRIPTION:
TMC207 is being investigated for the treatment of TB. TB is a contagious bacterial infection caused by M. tuberculosis that commonly affects the lungs, but can also affect other organs. Treatment of TB is protracted and burdensome and is further complicated by the emergence of multi-drug resistant M. tuberculosis strains. TMC207 is a diarylquinoline investigational compound that offers a novel mechanism of anti-TB action by specifically inhibiting mycobacterial adenosine triphosphate (ATP)-synthase. Multi-drug resistant TB (MDR-TB) is defined as infection with a strain of M. tuberculosis that is resistant to both INH and RMP (also known as rifampicin), two important drugs used to treat drug susceptible TB. Extensively drug-resistant TB (XDR-TB) is defined as MDR-TB with additional resistance to the most important second-line TB drugs, ie, one of the injectables (kanamycin, amikacin, or capreomycin) and fluoroquinolones. Pre-XDR TB is defined as MDR-TB with additional resistance to either a FQ or an injectable (kanamycin, amikacin, or capreomycin), but not to both a FQ and an injectable. Patients with either XDR-TB or pre-XDR will be included in this early access study. Patients who qualify for the study will be provided with a 24-week regimen of TMC207 which will be administered along with their background regimen (BR). BR drugs will be provided by the site investigator or designated study personnel in accordance with national TB program (NTP) guidelines. The BR should be constructed with at least 3 anti-tuberculosis drugs to which the patient's infection is known to be susceptible from recent drug susceptibility testing (DST) results (within the previous 6 months) or likely to be susceptible, based on known treatment history. The selection of the BR, including the number of companion drugs for TMC207, will be the responsibility of the investigator. At the screening visit, a completed inclusion/exclusion checklist list will be sent to the sponsor or its representative together with the patient's recent smear or culture and DST results (within preceding 6 months) and laboratory safety results to confirm eligibility. At baseline, a chest X-ray (CXR) will be taken in case no CXR or results of other imaging of the lungs are available within the previous month. Once treatment has been initiated, patients will be instructed to follow the visit schedule based on routine clinical care. Recommended visits and assessments should be planned 2, 4, 12, and 24 weeks following initiation of TMC207 in combination with the BR and 4 weeks (Week 28) and every 24 weeks (Weeks 48, 72, 96, and 120) after completion of TMC207 intake during the 96-week follow-up period. If needed, extra visits and assessments can be planned at the discretion of the investigator in order to best manage the patient's TB treatment. Patients who are taking clofazimine with TMC207 will require electrocardiogram (ECG) monitoring at mandatory protocol-specified visits. Serum chemistry (electrolytes) assessment will be performed at every visit in which an ECG is performed. After their last intake of TMC207, all patients will continue to take their BR under the supervision of their treating physician or local health center/hospital in accordance with NTP guidelines and local multi-drug resistant (MDR) TB treatment practice (i.e., treatment may be extended for reasons of complicated lung disease, etc.). Patients will be followed up for 96 weeks (2 years) after their last dose of TMC207 to evaluate the microbiological effect (verification of microbiological status [measured locally as per local standard of care; eg, smear, culture, DST] is recommended to be performed every 24 weeks) that TMC207 has provided these patients, as well as to monitor the safety and tolerability of TMC207. Patients who withdraw early, unless due to withdrawal of informed consent, will be followed for survival/clinical outcome (approximately every 6 months) until the early access study comes to an end in the patients' corresponding country. Patients can enter the study until TMC207 will be commercially available in the patient's country or can be accessed from another source or until discontinuation of the development program of TMC207.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pulmonary XDR or pre-XDR-TB infection with resistance to INH, RMP, and to a FQ and/or injectable second line TB drug (kanamycin, amikacin, or capreomycin). Confirmation should include previous (within the preceding 6 months) smear or culture and drug susceptibility testing (DST) results demonstrating pulmonary TB with an XDR or pre-XDR resistance pattern
* Patient has limited or no treatment options and is unable/ineligible to participate in any other TMC207 study
* Patient will be managed at a medical center that has been certified by the Green Light Committee of the World Health Organization (WHO) Stop TB Partnership, OR, following an assessment of the site confirms that the site meets equivalent standards. Patients must be able to receive at least 3 anti-TB drugs to which the patient's infection is known to be susceptible from recent DST results (within the previous 6 months) or likely to be susceptible, based on known treatment history, per availability in the country
* Patient is medically stable in the opinion of the investigator on the basis of physical examination, and safety examinations performed at screening
* Patients must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the early access study

Exclusion Criteria:

* History of and/or clinically relevant, currently active or underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, respiratory (other than due to TB), inflammatory, neoplastic, skin, immunological or infectious disease, which is not stable and controlled. If there are clinically relevant, currently active or underlying diseases, they should not compromise the safety of the patient or the ability to participate in the study as judged by the investigator. The investigator is encouraged to discuss concomitant illnesses with the sponsor
* Patients with complicated or severe extra-pulmonary manifestations of TB, including osteoarticular and central nervous system infection - Patients having received TMC207 in a previous study
* Any condition that, in the opinion of the investigator, would compromise the early access study or the well-being of the patient or prevent the patient from meeting or performing protocol requirements
* Current alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise patient's safety and/or compliance with the protocol procedures
* Patients with any clinically significant electrocardiogram abnormality at screening
* Patients having received medications (within the last 7 days prior to Day 1) that have the potential of prolonging the QT interval

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (5):
- Vilnius, Lithuania
- Russia (4):
  - Arkhangelsk
  - Moscow
  - Oryol
  - Saint Petersburg

REFERENCES:
- See also: Early Access of TMC207 in Combination With Other Anti-tuberculosis (TB) Drugs in Subjects With Extensively Drug Resistant (XDR) or Pre-XDR Pulmonary TB — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2427&filename=CR017233_CSR.pdf